CLINICAL TRIAL: NCT05647954
Title: A Randomized, Open-Label, Multicenter, Phase III Study of HX008 (a Humanized Monoclonal Antibody Against PD-1) Plus Transcatheter Arterial Chemoembolization (TACE) in the First-Line Treatment of Subjects With Stage IV (M1c) Melanoma That is Metastatic to the Liver
Brief Title: A Study of HX008 Plus Transcatheter Arterial Chemoembolization (TACE) in the First-Line Treatment of Subjects With Stage IV (M1c) Melanoma That is Metastatic to the Liver
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX008-Ⅲ-MM-01
Record Dates: First submitted 2022-11-28; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Melanoma Neuroendocrine Tumors Neuroectodermal Tumors Neoplasms Germ Cell and Embryonal Neoplasms by Histologic Type Neoplasms Neoplasms
MeSH Terms: interventions — Temozolomide; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HX008 Plus Transcatheter Arterial Chemoembolization(TACE) (Experimental)
  Interventions: Drug: HX008 + TACE
- Temozolomide Plus Transcatheter Arterial Chemoembolization (TACE) (Active Comparator)
  Interventions: Drug: Temozolomide + TACE
- Pembrolizumab (Active Comparator)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: HX008 + TACE — HX008 Subjects receive HX008 200 mg intravenous (IV) ,day1,every 3 weeks (Q3W) Procedure: TACE cisplatin 75 mg/sqm, day1, every 6 weeks; fotemustine 100 mg/sqm, day2, every 6 weeks; lipiodol is usually 5-10 ml (According to the location and number of lesions).
  Arms: HX008 Plus Transcatheter Arterial Chemoembolization(TACE)
Drug: Temozolomide + TACE — Temozolomide Subjects receive Temozolomide 200 mg/sqm intravenous (IV),day1-5, every 3 weeks (Q3W)
  Procedure: TACE :
  cisplatin 75 mg/sqm, day1, every 6 weeks; fotemustine 100 mg/sqm, day2, every 6 weeks; lipiodol is usually 5-10 ml (According to the location and number of lesions).
  Arms: Temozolomide Plus Transcatheter Arterial Chemoembolization (TACE)
Drug: Pembrolizumab — Subjects receive Pembrolizumab 2 mg/kg intravenous (IV),day1, every 3 weeks (Q3W)
  Arms: Pembrolizumab

SUMMARY:
The main purpose of this study is to compare the clinical benefit, as measured by Progression-Free Survival (PFS) and Overall Survival(OS), achieved by HX008 Plus Transcatheter Arterial Chemoembolization (TACE) or Temozolomide Plus Transcatheter Arterial Chemoembolization (TACE) in the First-Line Treatment of Subjects With Stage IV (M1c) Melanoma That is Metastatic to the Liver.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the Informed Consent Form（ICF）, understand the study, be willing to follow and be able to complete all test procedures;
2. Males or females, aged 18 to 75 are eligible on the day of signing the informed consent form;
3. Subjects with stage IV (M1c) melanoma confirmed by histology with liver metastasis approved by Pathology;
4. No prior systemic treatment for Stage IV (M1c) Melanoma with liver Metastatic; except:

   1. Melanoma with BRAF V600 mutation-positive may receive targeted therapy(e.g., BRAF/MEK inhibitor, alone or in combination) as first-line treatment for advanced or metastatic disease;
   2. Prior targeted therapy or immunotherapy (e.g., anti-PD-1 monoclonal antibody, anti-CTLA-4 monoclonal antibody or interferon, BRAF/MEK inhibitors, alone or in combination) as adjuvant or neoadjuvant therapy, if no recurrence or metastasis occurred during treatment or within 6 months of treatment termination. Prior adjuvant temozolomide and cisplatin chemotherapy of primary mucosa melanoma, without recurrence or metastasis during treatment or within 6 months of treatment termination.
5. Subjects must have a BRAF-V600 mutation or agree to carry out BRAF-V600 mutation detection during the screening phase ;
6. At least one measurable lesion of the subject's liver according to RECIST version 1.1 (Lesions with the longest diameter ≥ 10mm)
7. Target lesion has not received prior local treatment, including transarterial embolization (TAE), TACE, transarterial radioembolization (TARE), surgery, radiofrequency ablation (RFA), microwave ablation (MWA), other thermal ablation, percutaneous ethanol injection (PEI), radiation therapy, etc. Subjects who have received prior local treatment for non-target lesions are eligible for the study. Local treatment must be completed at least 4 weeks before randomization.
8. Liver function classified as Child-Pugh class A or B with a score ≤ 7, and no history of hepatic encephalopathy；
9. Suitability for the TACE procedures and chemotherapeutic agents pre-specified by the research center, without any contraindications;
10. Eastern Cooperative Oncology Group (ECOG) of 0 or 1;
11. Estimated life expectancy of ≥12 weeks;
12. Has sufficient organ and bone marrow function((no blood transfusions allowed for 14 days prior to blood routine, no any cell growth factors or/and platelet-raising drugs) to meet the following laboratory examination standards:

    1. Absolute neutrophil count (NUT#)≥1.5×10^9/L
    2. White blood cell count (WBC)≥3×10^9/L
    3. Platelet count (PLT)≥100×10^9/ L
    4. Hemoglobin (HGB)≥90 g/L

    f. Serum creatinine (Scr) ≤1.5×ULN g. ALT、AST ≤5×ULN h. TBIL≤1.5×ULN i.International normalized ratio (INR) ≤ 1.5×ULN; or activated partial thromboplastin time (APTT)≤ 1.5×ULN;(except for patients on anticoagulant therapy);
13. Women of childbearing age must have a negative pregnancy test within 72 hours before the first dose of trial treatment. Reproductive men and women of childbearing age are willing to take adequate contraceptive measures (e.g., oral contraceptives, intrauterine contraceptives, sexual abstinence or barrier contraceptives combined with spermicide) from signing the informed consent form to 12 months after the last administration of the trial drug;
14. The informed consent was voluntarily signed and the expected compliance was good.

Exclusion Criteria:

1. Malignant melanoma of ocular origin;
2. Investigator-identified contraindications to TACE (e.g., portal vein obstruction without formation of collateral vessels, etc.);
3. Liver lesions ≥ 10 cm in any dimension, more than 10 lesions on imaging evaluation, or liver lesions representing ≥ 50% of the liver volume.
4. Subjects diagnosed with any other malignancy within 3 years before randomization, except for malignancies with a low risk of metastasis and death (5-year survival rate > 90%), such as adequately basal cell or squamous cell skin cancer or carcinoma in situ of the cervix and other carcinomas in situ;
5. Had active autoimmune disease (except for psoriasis), that has required systemic treatment in the past 2 years((e.g., corticosteroids or immunosuppressive drugs). Except for alternative therapies (eg, thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency);
6. Need to receive systemic corticosteroids (dose equivalent to > 10 mg prednisone/day) or other immunosuppressive drugs within 14 days before enrollment or during the study period. Those under the following conditions are eligible:

   1. Locally external use or inhaled corticosteroids;
   2. short-term (≤7 days) use of glucocorticoids for the prevention or treatment of nonautoimmune allergic diseases;
7. Had received anti-tumor treatment within 4 weeks before randomization, or have not recovered from the toxicity of the last treatment (except for hair loss of Grade 2 and neurotoxicity of Grade 1);
8. Had received radiotherapy within 2 weeks before randomization， or had prior radiation therapy, or who has not recovered (≤ Grade 1 or at Baseline) from AEs due to previous radiation therapy;
9. Had received major surgery, open biopsy, or severe trauma within 4 weeks before randomization; Definition of major surgery: the minimum of 3 weeks of post-operative recovery time is required to undergo this study;
10. Had severe infection within 4 weeks or active infection requiring IV infusion or oral administration of antibiotics within 2 weeks before randomization;
11. Had participated in other drug or device clinical trials within 4 weeks before randomization;
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or found during the screening phase. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks, have no evidence of new or enlarging brain metastases, and also are off steroids 14 days before dosing with study medication may participate. Subjects with known untreated, asymptomatic brain metastases (ie, Lesions with numbers ≤ 3, and Lesions with the longest diameter ≤ 1 cm, ) may participate;
13. Has pleural effusion, pericardial effusion, or uncontrolled ascites requiring repeated drainage (once a month or more);
14. Has incomplete intestinal obstruction, active gastrointestinal bleeding, or perforation;
15. Has a history or current interstitial pneumonia, or current non--infectious pneumonitis treatment with corticosteroids;
16. Has uncontrolled cardiovascular disease, including but not limited to:

    1. heart failure greater than New York Heart Association (NYHA) class II
    2. unstable angina pectoris
    3. has myocardial infarction within 1 year
    4. supraventricular or ventricular arrhythmias with clinical significance poorly controlled without or despite clinical intervention;
17. Has uncontrolled systemic diseases, for instance, diabetes(Fasting Plasma Glucose ≥ 8.9 mmol/L or hypertension(systolic blood pressure ≥ 160 mmHg and / or diastolic blood pressure ≥ 100 mmHg);
18. Subjects with active tuberculosis;
19. History of human immunodeficiency virus infection, acquired or congenital immunodeficiency disease, organ transplantation, or stem cell transplantation;
20. Subjects with chronic hepatitis B or active hepatitis C. Except for Hepatitis B virus carriers or those with stable hepatitis B after drug treatment with DNA titer no higher than 500 IU/ml or copy number <2500 copies/ml, and cured hepatitis C patients (HCV RNA test negative);
21. Known to be allergic to macromolecular protein agents or monoclonal antibodies. Known to have a history of severe allergies to any of the chemotherapy drugs in the study ;
22. Alcohol dependence or drug abuse within the past 1 year;
23. Has received a live vaccine within 30 days before the first dose of trial treatment. Subjects are permitted to receive inactivated vaccines including those for seasonal influenza, intranasal influenza vaccines are not allowed;
24. Other reasons disqualifying the entering of this study are based on the investigators' evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) by Independent Review Committee(IRC) | 2 years
  PFS, defined as the time from randomization to the first documented disease.(HX008 + TACE vs Temozolomide + TACE)
Overall Survival (OS) | 2 years
  OS, defined as the duration from the start of treatment to death of any cause.(HX008 + TACE vs Temozolomide + TACE)

SECONDARY OUTCOMES:
Progression-free Survival (PFS) by Investigators | 2 years
  PFS, defined as the time from randomization to the first documented disease.(HX008 + TACE vs Temozolomide + TACE)
Objective Response Rate (ORR) | 2 years
  ORR, defined as the percentage of subjects achieving complete response (CR) and partial response (PR).
Disease Control Rate (DCR) | 2 years
  DCR, defined as the proportion of subjects achieving CR, PR, and Stable disease（SD) after treatment.
Duration of Response (DOR) | 2 years
  DOR, defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Progression-free Survival (PFS) by IRC or investigators | 2 years
  PFS, defined as the time from randomization to the first documented disease.(HX008 + TACE vs Pembrolizumab)
Overall Survival (OS) | 2 years
  OS, defined as the duration from the start of treatment to death of any cause.(HX008 + TACE vs Pembrolizumab)
Adverse events | 2 years
  Number of subjects with treatment-related adverse events as assessed by CTCAE v5.0,etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No